CLINICAL TRIAL: NCT04896125
Title: Comparison of Benzalkonium Chloride-containing Latanoprost and Preservative-free Bimatoprost on Ocular Surface Disease in Glaucoma Patients: a Prospective Randomised Study
Brief Title: Comparison of Different Drugs on Ocular Surface Disease in Glaucoma Patients: a Prospective Randomised Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201908054RINC
Record Dates: First submitted 2021-05-11; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2020-09

CONDITIONS: Glaucoma; Ocular Disorders (I.E. Caused by Ocular Disorders)
Keywords: Benzalkonium chloride; Ocular surface disease; Latanoprost; Bimatoprost
MeSH Terms: conditions — Glaucoma | interventions — Latanoprost

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lumigan PF: Patients older than 20 years were recruited from the Glaucoma Clinic of National Taiwan University Hospital. Patients were considered eligible for enrolment if they were newly diagnosed with glaucoma and started to receive ocular hypotensive eye drops at our clinic. Eligible patients then received 0.03% bimatoprost (preservative-free) (Lumigan PF, Allergan Inc., CA, USA).
  Interventions: Drug: Lumigan PF; Xalatan
- Xalatan: Patients older than 20 years were recruited from the Glaucoma Clinic of National Taiwan University Hospital. Patients were considered eligible for enrolment if they were newly diagnosed with glaucoma and started to receive ocular hypotensive eye drops at our clinic. Eligible patients then received 0.005% latanoprost (containing 0.02% BAK as a preservative) (Xalatan, Pfizer, NY, USA).
  Interventions: Drug: Lumigan PF; Xalatan
- Control: Patients older than 20 years were recruited from the Glaucoma Clinic of National Taiwan University Hospital. Patients were not diagnosed with glaucoma.

INTERVENTIONS:
Drug: Lumigan PF; Xalatan — Lumigan PF: 0.03% bimatoprost (preservative-free) Xalatan: 0.005% latanoprost (containing 0.02% BAK as a preservative) All patients were instructed to use only the given study medication during the study period.
  Groups: Lumigan PF; Xalatan

SUMMARY:
Participants were randomised to receive benzalkonium chloride-containing latanoprost (Xalatan) or preservative-free bimatoprost (Lumigan). Through this study, the investigators would like to analyze the impact of different antiglaucoma medications on ocular surface disease in glaucoma patients.

DETAILED DESCRIPTION:
The purpose of our study is to assess the effect of antiglaucoma medication on ocular surface disease in glaucoma patients before and after treatment with different antiglaucoma medication. All included patients are newly diagnosed with glaucoma and received no previous antiglaucoma treatment. Medical records will be collected prospectively from Sep. 15th 2019 to Aug. 31st 2022. The symptoms and signs of ocular surface disease in each individual will be assessed with questionnaire and clinical exams, including the basal Schirmer's test, non-invasive tear film breakup time, meibography, and in vivo confocal microscopy before and at 1, 3, 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients are not diagnosed with glaucoma and don't receive any ocular hypotensive eye drops at our clinic.
* Patients accept the rules for follow-up visits for at least six months.

Exclusion Criteria:

* Patients are with a history of ocular trauma.
* Patients are with contact lens use.
* Patients are diagnosed with secondary glaucoma.
* Patients have significant diseases affecting the meibomian gland and ocular surface.
* Patients have poor IOP control that required additional ocular hypotensive eye drops.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were considered eligible for enrolment if they were newly diagnosed with glaucoma and started to receive ocular hypotensive eye drops at our clinic.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
The influence of glaucoma eye drops on ocular surface disease index (OSDI) in patients | Change from Baseline OSDI at 1 month
The influence of glaucoma eye drops on ocular surface disease index (OSDI) in patients | Change from Baseline OSDI at 4 month

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan